CLINICAL TRIAL: NCT05972447
Title: Evaluation of Immediately Placed Ultra-wide Diameter Implant Placed in Mandibular Molars
Brief Title: Ultra-wide Diameter Implants in Mandibular Molars
Acronym: UWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdelrahman Elshahawy (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Elshahawy, principle investigator, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0210-01/2021
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Dental Implants
Keywords: UWD implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-restorable mandibular molar teeth (Other): patients with non restorable mandibular molar teeth without any periapical pathosis to be extracted and implanted immediately using ultrawide diameter dental implants
  Interventions: Procedure: Immediate implant placement of Ultrawide diameter dental implants

INTERVENTIONS:
Procedure: Immediate implant placement of Ultrawide diameter dental implants — immediate placement of ultrawide diameter dental implants in a fresh extraction socket of mandibular molar teeth
  Other Names: Ultrawide diameter dental implants

SUMMARY:
The goal of this [clinical trial] is to [To evaluate both the clinical and radiographical outcome on osteointegration and peri-implant bone density when using ultra wide diameter implant placed immediately in molar extraction socket]

DETAILED DESCRIPTION:
the aim of this study is to evaluate the clinical and radiographical outcomes on osseointegration and peri-implant bone density when using 12 ultrawide diameter dental implants placed immediately in 12 patients after atraumatic extraction of non-restorable mandibular molars without raising a flap or using bone grafts.

ELIGIBILITY:
Inclusion Criteria:

Adult patients ranging from 20-40 years.

* Adequate bone beyond teeth apices without jeopardizing any anatomical structure.
* Non-restorable mandibular molar teeth.
* Available bone with adequate width and buccolingual dimensions.
* Peri-implant bone defect should be 2mm or lesser.

Exclusion Criteria:

* Smokers.
* Medically compromised patients like uncontrolled diabetes and coagulation disorders.
* Tooth with periapical pathosis or bony defects.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
the mean value of implant stability | up to 6months
  The implant stability was measured by implant stability meter (Osstell™) immediately postoperative and at 6 months.
the mean value of peri-implant bone density | up to 9 months
  Radiographic evaluation of the bone density around each implant was done using OnDemand3D™.
the mean value of Marginal bone loss | up to 9months
  marginal bone levels were calculated from the reconstructed corrected sagittal views by drawing a line parallel to the implant serration extending from the crestal bone to the apical end of the implant. Average readings of the two sides at each interval were calculated and tabulated for statistical analysis.
the mean of peri-implant probing depth | up to 9 months
  Probing depth was assessed according to Gallagher and Silver Probing pocket depth refers to the distance between the gingival margin and the bottom of the pocket

CONTACTS AND LOCATIONS:
Overall Officials: Gaafar N Elhalawani, Study Director — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT05972447/Prot_SAP_000.pdf